CLINICAL TRIAL: NCT04105491
Title: Patient's Expectations, Preferences, Experiences Before, During and After the Treatment With Invisalign® Aligners
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Michael Nemec, Dr. med. dent Dr. med. univ, Medical University of Vienna
Other Study IDs: 1563/2019
Record Dates: First submitted 2019-09-04; First posted 2019-09-26 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Surveys and Questionnaires; Quality of Life; Orthodontics; Orthodontic Appliances

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Aligner Patients: Patients who decided to be treated with Invisalign® aligners
  Interventions: Device: IInvisalign® Aligners

INTERVENTIONS:
Device: IInvisalign® Aligners — Clear aligner orthodontic treatment

SUMMARY:
Orthodontic treatment extends over a longer period of time. lt takes months or rather years and it is no short-term treatment. The current literature does not answer the question of patients' expectations on aligner treatment and patients' experiences during aligner therapy sufficiently. Therefore, it is clinically and ethically highly relevant to know answers to these questions. This knowledge can highly improve the orthodontic consultation and therapy as well as the patients' comfort and wellbeing during the therapy. The proposed questionnaire-based interview survey is anticipated as a two-vear study.

In the first year study patients' expectations and preferences before the aligner treatment with Invisalign® aligners will be evaluated as well as preliminary changes in quality of life during the first stages of the Invisalign® aligner treatment. In the second year study it is planned to continue with the time equivalent questionnaires of the first year study and to investigate the patients' expectations, patients' experiences and levels of quality of life during and after aligner treatment. Therefore, it is planned to enroll 55 patients in this multicentre questionnaire-based interview survey. Two different questionnaires will be handed out to the patients. The first questionnaire, the aligner questionnaire, collects information from three different time points regarding the patients' expectations, preferences, experiences and views on second opinion concerning the aligner treatment. The results of those three time points, i.e. first (Ta0 before treatment begin), second (Ta6Mo, after 6 months of treatment) and third (Ta final, after finishing the treatment) will be statistically described and compared over time.

We expect most questionnaires of the second (during aligner treatment) and third time points (after finishing of treatment) to be evaluated by the end of the second year (second-year study), as the average treatment duration is about two years. The aim of the second questionnaire (OHlP 14) is to find out the changes in quality of life and is scheduled be started already in the firsfyear study. This questionnaire will be handed out to the patients before the treatment begins (Tq0), at the first check-up after the beginning of the treatment (TqCo1) and semi-annually afterwards (Tq6Mo' Tq12Mo, Tq18Mo, Tq24Mo, Tq30Mo) and finally at the end of the treatment (Tq final).

DETAILED DESCRIPTION:
It is planned to enroll 55 patients in this study, which is designed as a longterm questionnaire-based multicenter survey. Patients have to give their written consent prior to the study. Patients of the Clinical Division of Orthodontics at the University Clinic of Dentistry in Vienna as well as of a private practice will be included in order to increase the results' significance. All patients will be examined beforehand in order to exclude other pre-orthodontical treatment. After a short briefing about the aligner procedure and the therapeutic alternatives, each patient is selected for the aligner treatment with lnvisalign®. At this stage the chosen patient will be informed about the survey. The patient will receive the written consent form and the patient information form to think about at home. Should the patient consider to take part in the study, the signed forms must be returned at the following appointment. The patient will now receive the details about the different questionnaires and the estimated time per questionnaire (approximately 10 mins).

Before the first treatment the patient is asked to fill out the first OHIP G 14 (Tq 0) and the first aligner-questionnaire (Ta 0). The participants will be categorized by gender' age and level of education (compulsory school degree, higher school certificate, apprenticeship, university degree). Patients who have already been treated with aligners will not be included in the study. The routine-made initial and final scans of the patients will be evaluated according to the criteria of the orthodontic PAR (peer assessment rating) index. lnclusion criteria:

* Invisalign® "full" aligner treatment
* Invisalign® "lite" aligner treatment
* Adult patients (18 years and older)

Exclusion criteria:

* Previous aligner treatment
* Combined orthodontic and orthognathic surgical treatment
* Combined bracket and aligner treatment

The OHIP G 14 (Oral Health lmpact Profile G 14) questionnaire is an established and validated tool to evaluate the patients' quality of life. OHIP G 14 is the German version of OHIP (Oral Health lmpact Profile) 14. OHIP-14 is a short form of the oral health impact profile whose theoretic framework was based on a World Health Organization's International Classification of lmpairments, Disabilities and Handicaps relating health and its sequence in a hierarchy of different outcome levels. OHIP-14 has 7 conceptualized domains (2 items per domain): functional limitation, physical pain, psychological discomfort, physical disability, psychological disability, social disability and handicap. Patients are asked to rate how frequently they experienced an oral health impact (as described by each item). The response to each item is scored on a s-point Likert scale: 0, never; 1, hardly ever; 2, occasionally; 3, fairly often; and 4, very often or every day. Summary OHIP-14 scores can range from 0 to 56, and domain scores can range from o to 8. A higher oHlP-14 score indicates poorer oral health related quality of life (4-6) The OHIP questionnaire will be handed out to the patients before the treatment begins (Tq 0), at the first check-up after beginning of treatment (Tq Co1) - (usually 4 weeks after treatment) - and semi-annually afterwards (Tq6Mo, Tq12Mo' Tq18Mo' Tq24Mo, Tq3OMo) and at the end of treatment (Tq final). In order to simplify the questionnaires and spare pages, both questionnaires (OHIP G 14 and aligner questionnaire) will be merged into one questionnaire sheet, if applicable (at time points T0. T6 and Tfinal). Aligner-questionnaires will be handed out before (Ta0), after 6 months of treatment (Ta6) and at the end of treatment (Ta final). As there are no existing and comparable templates aiming at the study objectives, we designed the questionnaire according to a study on patients' perspectives on dental implant and bone graft surgery. lt is planned to explore how the patients' expectations change before, during and after treatment. Furthermore, each patient can evaluate his/her experiences with the aligner therapy after 6 months (most of the supportive procedures such as interproximal enamel reduction, wearing intermaxillary elastics, bonding of attachments will latest be started by then) and at the end of the treatment. The patients will be asked specific questions concerning aligner-treatment before, during and after the aligner-treatment.

Patients will get a reminder of the second and last aligner-questionnaire at one previous appointment. The estimated answer duration is going to be mentioned again' The patients are asked to fill out the third aligner-questionnaire on the day of the last appointment of active aligner therapy or within 8 weeks after the treatment Further, it is planned to correlate the patients' expectations concerning the treatment process/-success, their willingness for seeking a second opinion and their acceptance of different treatment modalities (interproximal enamel reduction, intermaxillary elastics) to the reported quality of life, the level of education, the grade of the PAR index at the beginning of treatment, as well as to gender and age.

The questionnaire will be arranged into the following sections:

1. Patient expectations will be asked at three different time points (before, during and after therapy) for their expectations at:
2. Patient experiences will be asked at two different time points (during and after therapy) concerning:
3. Patient preferences and acceptances will be asked at three different time points (before, during and after therapy) concerning:
4. Patient willingness to seek a second opinion will be explored at three different time points (before, during and after therapy) in consideration of:

Power calculations were done using the usual formulas for the paired t-test, adjusting for the planned use of non-parametric analysis by using the asymptotic relative efficiency (ARE). Assuming a SD (standard deviation) of 3.0 (from Liu 2011), a minimal sample size of 33 is needed to achieve a power of 0.95, to detect a clinically meaningful change of 2 in OHIP at significance level 0.05. Accounting fot 40% expected drop out due to the long-term character of the planned study, we arrive at a final sample size of 55 [33(1 - 0.4 dropout]. Due to the preliminary character of the questionnaire, there is no previous experience (clinical or otherwise) to base any sample size calculations on. Considering the fact that compared to the standardized and general OHIP, the questions in the new questionnaire are more detailed and tailored to the treatment these specific patients receive, we expect the power for this new questionnaire to be at least equal to the one computed for OHIP. Proportional odds mixed model will be used for OHIP questionnaires and for aggregate scores of aligner questionnaires, with covariate age, gender, level of education, reported quality of life and the grade of the PAR index at the beginning of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Invisalign® "full" aligner treatment
* Invisalign® "lite" aligner treatment
* Adult patients (18 years and older)

Exclusion Criteria:

* Previous aligner treatment
* Combined orthodontic and orthognathic surgical treatment
* Combined bracket and aligner treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who decided to be treated with Invisalign® aligners
Sampling Method: Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2019-09-16 (Actual); Primary Completion 2022-09-16 (Actual); Study Completion 2023-09-16 (Estimated)

PRIMARY OUTCOMES:
Patient expection on aligner therapy | up to 6 months
  before treatment has started

SECONDARY OUTCOMES:
Patient preferences and acceptences on aligner therapy | up to 12 months
  during treatment
Patient experiences on aligner therapy | up tp 24 months
  after aligner therapy

CONTACTS AND LOCATIONS:
Locations (1):
- University Dental Clinic Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Flores-Mir C, Brandelli J, Pacheco-Pereira C. Patient satisfaction and quality of life status after 2 treatment modalities: Invisalign and conventional fixed appliances. Am J Orthod Dentofacial Orthop. 2018 Nov;154(5):639-644. doi: 10.1016/j.ajodo.2018.01.013. PMID 30384934
- [Background] Pacheco-Pereira C, Brandelli J, Flores-Mir C. Patient satisfaction and quality of life changes after Invisalign treatment. Am J Orthod Dentofacial Orthop. 2018 Jun;153(6):834-841. doi: 10.1016/j.ajodo.2017.10.023. PMID 29853241
- [Background] Azaripour A, Weusmann J, Mahmoodi B, Peppas D, Gerhold-Ay A, Van Noorden CJ, Willershausen B. Braces versus Invisalign(R): gingival parameters and patients' satisfaction during treatment: a cross-sectional study. BMC Oral Health. 2015 Jun 24;15:69. doi: 10.1186/s12903-015-0060-4. PMID 26104387
- [Background] Liu Z, McGrath C, Hagg U. Changes in oral health-related quality of life during fixed orthodontic appliance therapy: an 18-month prospective longitudinal study. Am J Orthod Dentofacial Orthop. 2011 Feb;139(2):214-9. doi: 10.1016/j.ajodo.2009.08.029. PMID 21300250
- [Background] Slade GD, Spencer AJ. Development and evaluation of the Oral Health Impact Profile. Community Dent Health. 1994 Mar;11(1):3-11. PMID 8193981
- [Background] Slade GD. Derivation and validation of a short-form oral health impact profile. Community Dent Oral Epidemiol. 1997 Aug;25(4):284-90. doi: 10.1111/j.1600-0528.1997.tb00941.x. PMID 9332805